CLINICAL TRIAL: NCT04451928
Title: Prediction of Preterm Delivery by Serum Ischemia Modified Albumin, Biglycan and Decorin Levels in Women With Threatened Preterm Labour
Status: Completed | Type: Observational
Sponsor: Ismail Biyik (Other)
Responsible Party: Sponsor-Investigator, Ismail Biyik, Assistant Professor, Kutahya Health Sciences University
Organization: Kutahya Health Sciences University (Other)
Other Study IDs: 2020/01-1
Record Dates: First submitted 2020-06-25; First posted 2020-06-30 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Preterm Birth
Keywords: preterm birth; ischemia modified albumin; biglycan; decorin; prediction
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 13 Months
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Preterm delivery: Pregnant women who give birth before 37th gestational week
  Interventions: Diagnostic Test: Serum sample analysis
- Term delivery: Pregnant women who will give birth 37th and after gestational week
  Interventions: Diagnostic Test: Serum sample analysis

INTERVENTIONS:
Diagnostic Test: Serum sample analysis — Analysis of the levels of ischemia-modified albumin, biglycan and decorin levels

SUMMARY:
In this study, the levels of ischemia modified albumin, biglycan and decorin in the serums of pregnant women hospitalized for preterm labor will be examined. Their serum levels will be compared between women having preterm and term delivery. Their accuracy will be asessed in predicting preterm birth.

DETAILED DESCRIPTION:
The study will include 90 singleton pregnant women between the ages of 18 and 42 and gestational ages of 24 and 37 weeks.

Inclusion criteria:

* Singleton pregnancy
* Gestational age between 24 and 37 weeks
* Cervical dilatation less than 3 cm and cervical effacement less than 80%
* Uterine contraction ≥3 times at 30 minutes
* Intact amniotic membrane

Excusion criteria:

* Multiple pregnancy
* Preterm premature rupture of membranes
* Abnormal placentation (such as placenta previa)
* Uterin anomaly
* Maternal heart disease
* Inflammatory or infectious disease
* Preeclampsia
* Fetal growth restriction
* Congenital fetal anomaly
* Polyhydramnios
* Acute chorioamnionitis
* Medically induced preterm delivery

Patients who are hospitalized due to preterm labor will primarily receive bed rest and hydration. If cervical changes persist or if contractions continue after 2 hours after intravenous hydration, tocolytic treatment will be started. Calcium channel blockers will be used as tocolytic drug. Maternal corticosteroid (12 mg intramuscular betamethasone within 24 hours) will be given to accelerate fetal lung development. After 48 hours after steroid administration, tocolysis will be stopped. Demographic datas of the patients will be recorded. Patients will be followed until delivery. The gestational week will be determined according to the last menstrual date and will be confirmed by early ultrasonographic measurements. The gestational week at birth and the time between admission to the hospital and birth will be recorded. Delivery time will be divided into groups within 24 hours, 48 hours, 7 days, 14 days, and ≤37 weeks after admission. Mode of delivery, baby's birth weight, APGAR score will be recorded.

Venous blood samples will be taken from patients before medication. Serum samples will be stored in the cooler set to -80 °C until analysis. Levels of ischemia-modified albumin, biglycan and decorin levels will be examined by enzyme-linked immunosorbent assay (ELISA) method.

Statistical analysis:

After the assessment of the data, the variables between two groups will be compared by Mann Whitney U test, Student T test, Fisher Exact Test, Chi-Square Analysis. Regression model will be conducted in order to estimate the probability of the preterm birth. A value of p < 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Gestational age is between 24-37 weeks
* Cervical dilatation less than 3 cm and cervical effacement less than 80%
* Uterine contraction ≥3 times at 30 minutes
* Intact amniotic membrane

Exclusion Criteria:

* Multiple pregnancy
* Preterm premature rupture of membranes
* Abnormal placentation (such as placenta previa)
* Uterine anomaly
* Maternal heart disease
* Inflammatory or infectious disease
* Preeclampsia
* Fetal growth restriction
* Congenital fetal anomaly
* Polyhydramnios
* Acute chorioamnionitis
* Medically induced preterm delivery

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Singleton pregnant women between the ages of 18 and 42 and gestational ages of 24 and 37 weeks.
Study Population: Patients who are hospitalized due to preterm labor. Preterm labor is defined as regular contractions (uterine contraction ≥3 times at 30 minutes) of the uterus resulting in changes in the cervix that start before 37 weeks of pregnancy.
Sampling Method: Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-02-05 (Actual); Study Completion 2021-02-05 (Actual)

PRIMARY OUTCOMES:
Gestational age at birth | December 2019 - January 2021
  Preterm: <37 gestational week Term: ≥37 gestational week

SECONDARY OUTCOMES:
Hospital admission and delivery interval | December 2019 - January 2021
  Delivery time will be divided into groups within; 48 hours, 7 days, 14 days,
  * 35 weeks and
  * 37 weeks after hospital admission.
Mode of delivery | December 2019 - January 2021
  Vaginal delivery Cesarean delivery
APGAR score | December 2019 - January 2021
  Apgar stands for "Appearance, Pulse, Grimace, Activity, and Respiration." of newborn at 1 and 5 minutes after delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Ismail Biyik, MD, Principal Investigator — Kütahya Medical Sciences University
Locations (1):
- Kütahya Medical Sciences University, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rossi A, Bortolotti N, Vescovo S, Romanello I, Forzano L, Londero AP, Ambrosini G, Marchesoni D, Curcio F. Ischemia-modified albumin in pregnancy. Eur J Obstet Gynecol Reprod Biol. 2013 Oct;170(2):348-51. doi: 10.1016/j.ejogrb.2013.06.037. Epub 2013 Jul 23. PMID 23891063
- [Background] Underhill LA, Avalos N, Tucker R, Zhang Z, Messerlian G, Lechner B. Serum Decorin and Biglycan as Potential Biomarkers to Predict PPROM in Early Gestation. Reprod Sci. 2019 Mar 21:1933719119831790. doi: 10.1177/1933719119831790. Online ahead of print. PMID 30895897
- [Derived] Biyik I, Soysal C, Ince OUO, Durmus S, Oztas E, Keskin N, Isiklar OO, Karaagac OH, Gelisgen R, Uzun H. Prediction of Preterm Delivery Using Serum Ischemia Modified Albumin, Biglycan, and Decorin Levels in Women with Threatened Preterm Labor. Rev Bras Ginecol Obstet. 2023 Dec;45(12):e754-e763. doi: 10.1055/s-0043-1772593. Epub 2023 Dec 23. PMID 38141595